CLINICAL TRIAL: NCT03301168
Title: Phase I/II Study of CaspaCIDe® T Cells From an HLA-Partially Matched Family Donor After Negative Selection of TCR αβ+T Cells in Pediatric Patients Affected by Hematological Disorders
Brief Title: Study of Gene Modified Donor T-cells Following TCR Alpha Beta Positive Depleted Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-U-004
Expanded Access: NCT03639844 (No longer available)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia, Acute Myeloid (AML), Child; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Primary Immune Deficiency Disorder; Osteopetrosis; Cytopenia; Hemoglobinopathy in Children; Anemia, Aplastic
Keywords: ALL; AML; hematologic neoplasms; hematologic malignancies; primary immune deficiences; allogeneic stem cell transplant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Primary Immunodeficiency Diseases; Osteopetrosis; Cytopenia; Anemia, Aplastic; Hematologic Neoplasms | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BPX-501 T cells and Rimiducid (Experimental): TCR alpha beta depleted graft infusion with addback of BPX-501 T cells.
  Rimiducid: Dimerizer drug administered to subjects who present with Grade I-IV acute GVHD with inadequate response to steroids within 48 hours of treatment or mild to severe chronic GVHD with inadequate response to steroids within 7 days of treatment.
  Interventions: Biological: BPX-501 T cells; Drug: Rimiducid

INTERVENTIONS:
Biological: BPX-501 T cells — T cells transduced with CaspaCIDe® safety switch
  Other Names: rivogenlecleucel
Drug: Rimiducid — administered to inactivate BPX-501 cells in the event of GVHD
  Other Names: AP1903

SUMMARY:
This study will evaluate pediatric patients with malignant or non-malignant blood cell disorders who are having a blood stem cell transplant depleted of T cell receptor (TCR) alfa and beta cells that comes from a partially matched family donor. The study will assess whether immune cells, called T cells, from the family donor, that are specially grown in the laboratory and given back to the patient along with the stem cell transplant can help the immune system recover faster after transplant. As a safety measure these T cells have been programmed with a self-destruct switch so that they can be destroyed if they start to react against tissues (graft versus host disease).

DETAILED DESCRIPTION:
This is a Phase 1/2 study evaluating the safety and feasibility of BPX-501 T cells infused after partially mismatched, related, TCR alpha beta T cell depleted hematopoietic stem cell transplant (HSCT) in pediatric patients. The purpose of this clinical trial is to determine whether BPX-501 infusion can enhance immune reconstitution in those patients with hematologic disorders, with the potential for reducing the severity and duration severe acute graft versus host disease (GvHD).

The trial will also evaluate the treatment of GvHD by the infusion of dimerizer drug (AP1903/rimiducid) in those subjects who present with GVHD that does not adequately respond to standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 1 month and < 26 years
2. Life expectancy > 10 weeks
3. Subjects deemed eligible for allogeneic stem cell transplantation.
4. Subjects with life-threatening hematological malignancies (high-risk ALL in 1st CR, ALL in 2nd or subsequent CR, AML in 1st CR, AML in 2nd or subsequent CR, myelodysplastic syndromes, non-Hodgkin lymphomas in 2nd or subsequent CR, other hematologic malignancies eligible for stem cell transplantation per institutional standard);
5. Non-malignant disorders amenable to cure by an allograft:

   1. primary immune deficiencies,
   2. severe aplastic anemia not responding to immune suppressive therapy,
   3. osteopetrosis,
   4. hemoglobinopathies, (thalassemias, and sickle cell anemia, and Diamond-Blackfan anemia among others)
   5. congenital/hereditary cytopenia, including Fanconi Anemia before any clonal malignant evolution (MDS, AML) Note: Subjects will be eligible if they meet either item 4 OR item 5.
6. Lack of suitable conventional donor (HLA identical sibling or HLA phenotypically identical relative or 10/10 unrelated donor evaluated using high resolution molecular typing) or presence of rapidly progressive disease not permitting time to identify an unrelated donor
7. A minimum genotypic identical match of 5/ 10 is required.
8. The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA- DRB1 and HLA-DQB1.
9. Lansky/Karnofsky score > 50
10. Signed written informed consent

Exclusion Criteria:

1. Greater than Grade II acute GVHD or chronic extensive GVHD due to a previous allograft at the time of inclusion
2. Subject receiving an immunosuppressive treatment for GVHD treatment due to a previous allograft at the time of inclusion
3. Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance < 30 mL / min)
4. Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction < 40%)
5. Current active infectious disease (including positive HIV serology or viral RNA)
6. Serious concurrent uncontrolled medical disorder
7. Pregnant or breastfeeding subject
8. For subjects who have received more than 1 x 10E5 alpha/beta T cells/kg with the graft infusion the clinical trial site must contact the sponsor for approval to be eligible to receive BPX-501 infusion.

Ages: 1 Month to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Month 24
  Demonstrate safety of BPX-501 MTD
TRM/NRM | Day 180, Month 12
  Assess the cumulative incidence of non-relapse/transplant related mortality

SECONDARY OUTCOMES:
Disease-free survival | Month 24
  Disease-free survival rates after transplantation
Relapse | Month 12
  Cumulative incidence of relapse
Engraftment | Month 24
  Cumulative incidence of neutrophil and platelet engraftment, primary & secondary graft failure
GvHD | Month 24
  Cumulative incidence and severity of acute and chronic GvHD
Rimiducid Efficacy | Month 24
  Time to resolution of acute or chronic GvHD after administration of rimiducid
Infection | Month 24
  Rate of infectious complications
Hospitalizations | Month 24
  Duration of hospitalization and rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University - Division of Pediatric Stem Cell Transplant & Regenerative Medicine, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Dana-Farber Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts
  - Children's Hospital at Montefiore, The Bronx, New York
  - Oregon Health Sciences University - Doernbecher Children's Hospital, Portland, Oregon
  - University of Texas Southwestern-Children's Medical Center, Dallas, Texas
  - Baylor College of Medicine/ Texas Children's Hospital, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No